CLINICAL TRIAL: NCT00321412
Title: A Double-blind, Randomized, Placebo-controlled Multicenter Study to Assess the Safety and Efficacy of AST-120 in Mild to Moderately Active Crohn's Patients With Fistulas
Brief Title: Safety and Efficacy of AST-120 in Mild to Moderate Crohn's Patients With Fistulas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocera Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AST001
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Inflammatory Bowel Disease; Intestinal Fistula
Keywords: Crohn's disease; IBD; Inflammatory Bowel Disease; Fistula
MeSH Terms: conditions — Inflammatory Bowel Diseases; Intestinal Fistula; Crohn Disease; Fistula | interventions — AST 120

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Celphere® CP-305, stained to match appearance of AST-120, in 2g sachets
  Interventions: Drug: AST-120
- 1 (Experimental): AST-120, 2 gram sachets
  Interventions: Drug: AST-120

INTERVENTIONS:
Drug: AST-120 — oral, sachet, 2 grams three times daily for 8 weeks

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the experimental drug AST-120 in treating patients with mild to moderately severe Crohn's disease who have fistulas. The study will test whether or not patients receiving AST-120 experience a greater reduction in number of draining fistulas and improvement of their other Crohn's disease symptoms versus patients who receive placebo (material that does not contain any active medication).

DETAILED DESCRIPTION:
The experimental drug AST-120 is composed of black, odorless spherical carbon particles in 2g sachets (aluminum foil pouches). The placebo consists of microcrystalline cellulose spheres, Celphere CP-305, stained to match the appearance of AST-120, in 2g sachets (aluminum foil pouches). Both AST-120 and placebo are oral (taken by mouth)preparations. Both are tasteless. To take the product, patients will tear open the sachets, drop the contents directly on their tongue and wash it down with 8 ounces of water.

Patients will be randomly assigned (like the toss of a coin), to receive either AST-120 or placebo. Patients will have a 50/50 chance of receiving placebo. Patients who participate in this study will be required to take a single dose of study drug (AST-120 or placebo) 3 times a day, 30 minutes after a meal, for 8 weeks, and be evaluated at Week 4 and Week 8. This is a 'blinded' treatment, which means that neither the patient nor the study doctor will know if the patient has received study drug or placebo.

If, at the end of the first full course of randomized treatment, (8 weeks), patients are not showing an improvement in their condition, they may have the option to receive the alternate blinded treatment for one treatment course (8 weeks). The study doctor will discuss this option with each patient individually. During this second course of treatment, patients will be evaluated at Week 12 and Week 16. If the patient does not respond to the alternate blinded treatment, or their condition worsens after 4 weeks (assessed at Week 12), they may be removed from the study at the discretion of the investigator.

If patients respond to either the initial treatment or the alternate blinded treatment, they will have monthly doctor/clinic visits for up to 6 months (Week 24), or until their condition worsens or they relapse. Patients will not receive any study drug during this follow-up period.

Relapse is defined for this study as:

* an increase by 1 or more in the number of draining fistulas for 2 sequential visits versus the number present at the time of response (response is defined as at least a 50% reduction in the number of draining fistulas at either Week 8, or for those patients receiving alternate blinded treatment, Week 16).

There are a maximum of 8 patient evaluation visits in this study (Screen, Baseline, Week 4, Week 8, Week 12, Week 16, Week 20 and Week 24). Evaluations at most of these visits include a review of concomitant medications, medical history/adverse events, physical exam, fistula exam, blood draws for safety labs, urine pregnancy tests for females, and measurement of body weight. Patients will also be asked to keep a daily diary to record frequency of bowel movements, general well-being, and use of antidiarrheal medication.

Treatment failure in this study is defined by one or more of the following occurring prior to Week 8:

* The need for additional therapies or dose increase for treatment of Crohn's disease, including an increase of corticosteroid dose to higher than baseline
* Clinical/symptomatic development of an abscess
* Clinical/symptomatic evidence of stricture
* The need for surgical intervention for Crohn's disease
* The patient withdraws from the study

Patients will be discontinued from the study at any time if one or more of the following complications occur:

* Development of an abscess or symptomatic stricture
* The need for surgical intervention for Crohn's disease
* Occurrence of any other event that in the opinion of the investigator warrants discontinuation of the patient from the study

In addition, patients whose CDAI score has risen by > or = 70 points above baseline or risen above 400 will be discontinued from the study.

Administration of any additional therapies or dose increases of concomitant medications (including corticosteroids) to control Crohn's disease to higher than baseline while receiving study drug (initial randomized treatment or alternate blinded treatment) will require discontinuation of the patient from the study.

Discontinued patients will be evaluated in a termination visit to document the lack of treatment efficacy and no further study treatment will be given.

ELIGIBILITY:
Inclusion Criteria:

* Body Weight > or = 40kg
* Documented diagnosis of Crohn's disease, including patients with documented diagnosis of ileitis, colitis, or ileocolitis
* Presence of at least one draining fistula. Patients with enterocutaneous fistulas can be included if they have > or = 1 draining perianal fistula. Women with rectovaginal fistulas can be included if they have > or = 1 draining perianal fistula.
* Crohn's Disease Activity Index (CDAI) score < 400
* Platelet count (thrombocytes) > or = 100,000/uL
* Able and willing to comply with all protocol procedures for the duration of the study
* Able and willing to understand, sign and date an informed consent document, and authorize access to protected health information
* Females must be postmenopausal, surgically incapable of bearing children, or practicing a reliable method of birth control (hormonal contraceptives, intrauterine devices, spermicide and barrier). Partner/spouse sterility may also qualify at the Investigator's discretion. Females of child-bearing potential must have a negative urine pregnancy test at baseline.

Exclusion Criteria:

* Non-response to infliximab or other biological immunosuppressants/ immunomodulators for fistulas associated with Crohn's disease (response is defined as a > or = 50% reduction from baseline in the number of fistulas over at least four weeks); patients who respond once to infliximab and eventually fail can be included
* Infliximab (and/or other biological immunosuppressant/immunomodulatory) therapy within 3 months prior to enrollment in the study
* Presence of symptomatic strictures or suggestion of significant clinical obstruction
* Patients with setons are excluded, unless the setons are removed within 48 hours prior to study entry
* Presence of entero-entero, recto-vesicular, entero-vesicular fistulas
* Platelet count (thrombocytes) < 100,000/uL
* CDAI score of > or = 400
* Patient is unable to stay on a stable dose of concomitant Crohn's disease medication(s) for at least 10 weeks in the opinion of the investigator
* Currently symptomatic untreated diarrhea due to conditions other than mild to moderately active Crohn's disease (e.g., bacterial or parasitic gastroenteritis, bile salt diarrhea, etc.)
* Severe diarrhea defined by > 10 liquid bowel movements per day
* Other local manifestations of mild to moderately active Crohn's disease such as abscesses, or other disease manifestations for which surgery might be indicated or which might preclude utilization of a CDAI to assess response to therapy (e.g., short bowel syndrome)
* Presence of an ileostomy
* Receiving Total Parenteral Nutrition (TPN) as the sole source of nutrition within 3 weeks of Screen
* Poor tolerability of venipuncture or lack of adequate venous access for required blood sampling.
* Hemoglobin < 8.5 g/dL (females) or hemoglobin < 10 g/dL (males) at Screen
* Women who are pregnant, breast feeding, or planning to become pregnant during the study
* Other major physical or major psychiatric illness within the last 6 months that in the opinion of the investigator would affect the patient's ability to complete the trial
* Uncontrolled systemic disease
* Patients undergoing chemotherapy for the treatment of cancer
* Known hypersensitivity or contraindication to any component of the test product (study drugs) or diagnostics used
* Participation in another study within eight (8) weeks prior to the study
* Unable to attend all visits required by the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Efficacy: The proportion of patients considered to be "treatment successes" defined by a reduction of at least 50% in the number of draining fistulas at both week 4 and week 8 of an 8 week treatment period | 8 weeks
Safety: Adverse events deemed possibly, probably or definitely related to study drug during 8 weeks of treatment | 8 weeks

SECONDARY OUTCOMES:
Efficacy: 100% non-draining fistulas at both week 4 and week 8 | 8 weeks
Efficacy: Fistula response at Week 8 | 8 weeks
Efficacy: Change in CDAI scores from baseline over 8 weeks of treatment | 8 weeks
Safety: Clinical laboratory tests (electrolytes) | 8 weeks
Safety: Development of abscesses | 8 weeks
Safety: Physical examination, vital signs (blood pressure, heart rate, respiration rate and temperature) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Fischer, MD, Study Director — Ocera Therapeutics
Locations (87):
- United States (25):
  - Advanced Clinical Research Institute, Anaheim, California
  - Digestive Care Medical Center, San Carlos, California
  - Shafran Gasteroenterology Center, Winter Park, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University, Outpatient Clinical Research Facility, Indianapolis, Indiana
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University of Louisville, Department of Surgery, Louisville, Kentucky
  - Metropolitan Gastroenterology Group/Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Drs. Scherf, Chessler, Zingler & Spinnell, MD, PA, Fort Lee, New Jersey
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Mount Sinai School of Medicine, IBD Research Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolina Digestive Health Associates, Charlotte, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic - Department of Gastroenterology, Cleveland, Ohio
  - The Penn State University, Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Digestive Disease Center/MUSC, Charleston, South Carolina
  - Memphis Gastroenterology Group, PC, Germantown, Tennessee
  - University of Washington, Seattle, Washington
  - Dean Foundation Research Center, Madison, Wisconsin
- Austria (3):
  - Univ Klinik fur Innere Medizin Innsbruck, Innsbruck
  - Universitatsklinik fur Innere Medizin I der PMU, Salzburg
  - AKH Wien - Univ Klinik Innere Med IV, Vienna
- Belgium (4):
  - Imelda General Hospital, Bonheiden
  - St. Jansziekenhuis/Ziekenhuis Oost-Limburg, Genk
  - University Hospital Gasthuisberg, University of Leuven, Leuven
  - H.-Hartziekenhuis Roeselare-Menen vzw, Roeselare
- Canada (5):
  - GILDR Group, University of Edmonton, Edmonton, Alberta
  - Liver & Intestinal Research Centre, Vancouver, British Columbia
  - McMaster University Medical Centre, Hamilton, Ontario
  - London Health Sciences Center, London, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Czechia (5):
  - University Hospital Brno, Internal and Gastroenterology Department, Brno
  - Regional Hospital Liberec, Department of Gastroenterology, Liberec
  - University Hospital Prague 2, 4th Department of Internal Medicine, Prague
  - Thomayer's University Hospital Prague, 2nd Internal Department, Prague
  - Institute for Clinical and Experimental Medicine, Prague
- France (9):
  - CHU Hopital Nord, Service de Gastro-enterologie et nutrition, Amiens
  - Hopital de la Cote de Nacre - CHU, Caen
  - CHU de Grenoble - Hopital Nord, Grenoble
  - Hopital Claude Huriez, Service des maladies de l'appareil disgestif, Lille
  - Hopital Nord, Service de Gastro-Enterologie, Marseille
  - Hopital Saint-Eloi, Service de Gastro-enterologie et transplantation, Montpelier
  - CHU Hotel Dieu, Institut des Maladies de l'Appareil Digestif, Nantes
  - CHU de Nice - Hopital de l'Archet 2, Nice
  - Hopital Leopold Bellan, Paris
- Germany (11):
  - Universitatsklinikum Aachen, Aachen
  - Charite-Campus Virchow-Klinikum, Berlin
  - Klinikum der Johann-Wolfgang-Goethe Universitat Frankfurt am Main, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinik Heidelberg Abteilung Gastroenterologie und Hepatologie, Heidelberg
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - Klinikum rechts der Isar der TUM II, München
  - Universitatsklinikum Regensburg, Regensburg
  - Universitat Rostock - Midizinische Fakultat, Rostock
  - Medizinische Universitatsklinik Tubingen, Tübingen
  - Universitatsklinikum Ulm, Ulm
- Hungary (4):
  - Peterfy Sandor utcai Korhaz-Rendelointezet, Budapest
  - Semmelweis Egyetem, Budapest
  - Miskolc Megyei Jogu Onkormanyzat Semmelweis Oktato Korhaz-Rendelointezet, Miskolc
  - Szegedi Tudomanyegyetem, I.sz. Belgyogyaszati Klinika, Szeged
- Israel (7):
  - Bnai Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Strauss Medical Center, Jerusalem
  - Meir Hospital, Kfar Saba
  - Rabin Medical Center, Bellinson Hospital, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
- Erasmus MC, Department of Gastroenterology and Hepatology, Rotterdam, Netherlands
- Poland (7):
  - Samodzielny Publiczny Centralny Szpital Kliniczny Slaskiej AM, Katowice
  - Zakaznych Szpitala Uniwersyteckiego w Krakowie, Krakow
  - Korektalnej Uniwersytetu Medycznego w Lodzi, Lodz
  - University Hospital Olomouc, 2nd Internal Department, Olomouc
  - Samodzielny Publiczny Szpital Kliniczny Nr 2 im. Heliodora, Poznan
  - Samodzielny Publiczny Centralny Szpital, Warsaw
  - Katedra Klinika Gastroenterologi, Akedemil Medycanej we Wroclawiu, Wroclaw
- United Kingdom (6):
  - Bristol Royal Infirmary, Dept. of Gastroenterology, Bristol
  - Countess of Chester Hospital, Chester
  - Crosshouse Hospital, Kilmarnock
  - Leicester General Hospital - GI Research Unit, Leicester
  - University College London Hospital, Dept. of Gastroenterology, London
  - John Radcliffe Hospital, Dept. of Gastroenterology, Oxford

REFERENCES:
- [Background] Hay JW, Hay AR. Inflammatory bowel disease: costs-of-illness. J Clin Gastroenterol. 1992 Jun;14(4):309-17. doi: 10.1097/00004836-199206000-00009. PMID 1607607
- [Background] Hugot JP, Chamaillard M, Zouali H, Lesage S, Cezard JP, Belaiche J, Almer S, Tysk C, O'Morain CA, Gassull M, Binder V, Finkel Y, Cortot A, Modigliani R, Laurent-Puig P, Gower-Rousseau C, Macry J, Colombel JF, Sahbatou M, Thomas G. Association of NOD2 leucine-rich repeat variants with susceptibility to Crohn's disease. Nature. 2001 May 31;411(6837):599-603. doi: 10.1038/35079107. PMID 11385576
- [Background] Ogura Y, Bonen DK, Inohara N, Nicolae DL, Chen FF, Ramos R, Britton H, Moran T, Karaliuskas R, Duerr RH, Achkar JP, Brant SR, Bayless TM, Kirschner BS, Hanauer SB, Nunez G, Cho JH. A frameshift mutation in NOD2 associated with susceptibility to Crohn's disease. Nature. 2001 May 31;411(6837):603-6. doi: 10.1038/35079114. PMID 11385577
- [Background] Best WR, Becktel JM, Singleton JW. Rederived values of the eight coefficients of the Crohn's Disease Activity Index (CDAI). Gastroenterology. 1979 Oct;77(4 Pt 2):843-6. PMID 467941
- [Background] Schwartz DA, Loftus EV Jr, Tremaine WJ, Panaccione R, Harmsen WS, Zinsmeister AR, Sandborn WJ. The natural history of fistulizing Crohn's disease in Olmsted County, Minnesota. Gastroenterology. 2002 Apr;122(4):875-80. doi: 10.1053/gast.2002.32362. PMID 11910338
- [Background] Hellers G, Bergstrand O, Ewerth S, Holmstrom B. Occurrence and outcome after primary treatment of anal fistulae in Crohn's disease. Gut. 1980 Jun;21(6):525-7. doi: 10.1136/gut.21.6.525. PMID 7429313
- [Background] Farmer RG, Hawk WA, Turnbull RB Jr. Clinical patterns in Crohn's disease: a statistical study of 615 cases. Gastroenterology. 1975 Apr;68(4 Pt 1):627-35. No abstract available. PMID 1123132
- [Background] Gray BK, Lockhartmummery HE, Morson BC. Crohn's disease of the anal region. Gut. 1965 Dec;6(6):515-24. doi: 10.1136/gut.6.6.515. No abstract available. PMID 5857889
- [Background] Schwartz DA, Pemberton JH, Sandborn WJ. Diagnosis and treatment of perianal fistulas in Crohn disease. Ann Intern Med. 2001 Nov 20;135(10):906-18. doi: 10.7326/0003-4819-135-10-200111200-00011. PMID 11712881
- [Background] Schwartz DA, Herdman CR. Review article: The medical treatment of Crohn's perianal fistulas. Aliment Pharmacol Ther. 2004 May 1;19(9):953-67. doi: 10.1111/j.1365-2036.2004.01917.x. PMID 15113362
- [Background] Present DH, Rutgeerts P, Targan S, Hanauer SB, Mayer L, van Hogezand RA, Podolsky DK, Sands BE, Braakman T, DeWoody KL, Schaible TF, van Deventer SJ. Infliximab for the treatment of fistulas in patients with Crohn's disease. N Engl J Med. 1999 May 6;340(18):1398-405. doi: 10.1056/NEJM199905063401804. PMID 10228190
- [Background] Present DH, Korelitz BI, Wisch N, Glass JL, Sachar DB, Pasternack BS. Treatment of Crohn's disease with 6-mercaptopurine. A long-term, randomized, double-blind study. N Engl J Med. 1980 May 1;302(18):981-7. doi: 10.1056/NEJM198005013021801. PMID 6102739
- [Background] Hanauer SB, Feagan BG, Lichtenstein GR, Mayer LF, Schreiber S, Colombel JF, Rachmilewitz D, Wolf DC, Olson A, Bao W, Rutgeerts P; ACCENT I Study Group. Maintenance infliximab for Crohn's disease: the ACCENT I randomised trial. Lancet. 2002 May 4;359(9317):1541-9. doi: 10.1016/S0140-6736(02)08512-4. PMID 12047962
- [Background] Sands BE, Anderson FH, Bernstein CN, Chey WY, Feagan BG, Fedorak RN, Kamm MA, Korzenik JR, Lashner BA, Onken JE, Rachmilewitz D, Rutgeerts P, Wild G, Wolf DC, Marsters PA, Travers SB, Blank MA, van Deventer SJ. Infliximab maintenance therapy for fistulizing Crohn's disease. N Engl J Med. 2004 Feb 26;350(9):876-85. doi: 10.1056/NEJMoa030815. PMID 14985485